CLINICAL TRIAL: NCT06618768
Title: Preventive Effect of Aronia Mixture Against UTI - a Pilot Study
Brief Title: Can Consumption of an Aronia-mixture Prevent Urinary Tract Infections in Female Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Collaborators: Ullevaal University Hospital (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Principal Investigator, Tonje Holte Stea, Professor, University of Agder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 422796 (REK)
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Urinary Tract Infection (Diagnosis)
Keywords: clinical trial; primary care; urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consumption of an aronia-mixture (Experimental): Participants will daily consume 1 dL aronia-mixture for 6 months. The mixture may be consumed in smaller portions throughout the day, but according to results from a non-clinical pilot-study (https://pubmed.ncbi.nlm.nih.gov/25026919/), the mixture should be consumed with a meal in order to avoid nausea. The aronia-mixture has been developed by the research group and produced for free by Ronia AS, Randaberg, Norway. The mixture is produced from aronia-berries (50%) and apples (50%), and 1 dL (one serving) consists of 600 mg proanthocyanidins, 300 mg anthocyanins and 100 mg chlorogenic acids with pH 3.6. Urine samples (25 mL) will be delivered at general practices for chemical analysis of metabolites from the intervention drink at day 0, 60, 120, and 180 (spot urine). In addition, an urine sample will be collected at day 0 for microbiological analysis (urine culture). The intervention will not replace any medical treatment during the project period.
  Interventions: Dietary Supplement: Consumption of an aronia-mixture to prevent Urinary Tract Infections in female patients

INTERVENTIONS:
Dietary Supplement: Consumption of an aronia-mixture to prevent Urinary Tract Infections in female patients — The present pilot study will assess the feasibility of methods and procedures to be used in a larger study and contribute to establish power calculations required to conduct a randomised clinical trial which will examine whether consumption of 1 dL aronia-mixture/day for six months will reduce prevalence of symptomativ UTi episodes among adult women with a recent history of uncomplicated, recurrent UTIs.

SUMMARY:
The goal is to determine the feasibility of conducting a randomised clinical trial to measure the effectiveness of an aronia mixture in reducing recurrence of urinary tract infections (UTIs) and antibiotic use by women with a history of frequent UTIs. In addition, the study aim to collect data in order to establish power calculations required for a full-scale study.

DETAILED DESCRIPTION:
Aronia berries have been and are used as a food, especially in Eastern Europe and the USA. No negative health effects have been reported from consuming similar amounts of aronia berries as those given to participants in this pilot study. On the contrary, studies suggest that consuming aronia berries has several positive health effects (1). The present 6-months pilot study will examine the feasibility of the study (recruitment process, drop-outs, program adherence, treatment duration, program accetability), identify potential biomarkers of the aronia-mixture and provide information to establish power calculations in a full-scale randomized controlled trial.

Outcomes in the pilot study is number of UTI episodes (both treated and untreated) corresponding to historical episodes (last 12 months), characterization of uropathogens from urine culture analyses, as well as characterization of phenolic metabolites in urine as a result of the intervention. Findings of catabolites based on certain polyphenols will reflect the intestinal ability to metabolize compounds (e.g. condensed tannins), and how these catabolites are absorbed into the circulatory system. Changes in the catabolite pattern will form the basis for estimation of the intervention period needed when planning a full-scale randomized controlled trial.

Research Team:

Tonje H Stea (Professor, University of Agder) - Project Leader Rune Slimestad (Chemist, PhD PlantChem AS) - Responsible for metabolite analysis of urine. Will provide intervention drink and urine containers to the medical office.

Nils Grude (Senior Physician, PhD Antibiotic Center, Ullevål Hospital) - Responsible for microbiology expertise.

Ståle Tofteland (Senior Physician, PhD, Kristiansand Hospital) - Responsible for cultivation and characterization of bacteria in urine.

Tor Jakob Rørvik (General Practitioner, Konsmo) - Responsible for participant approval and reception of urine samples.

Development of an aronia mixture (intervention drink) A mixture has been developed consisting of aronia and apple juices (1:1 ratio), and the mixture is concentrated by removing 50% of the liquid content in the form of water. Study participants will therefore consume a larger proportion of potential bioactive compounds than the proportion of bioactive compounds available in the equivalent volume of natural aronia juice. Apple juice has been added to the mixture in order to created a sweeter, more desirable flavor.

The mixture is thoroughly characterized in terms of ingredients, and a daily dose of 1 g of polyphenols will provide 680 mg of B-type proanthocyanidins, 125 mg of anthocyanins, and 215 mg of phenolic acids per dL aronia mixture.

Estimation of daily dose of aronia-mixture in the present study is based on the content of B-type proanthocyanidins, as metabolites of these compounds can provide a natural antibiotic effect on uropathogens. Specifically, the dosage used in this study has been calculated based on a previous pharmacokinetic study among students at the Univeristy of Oslo (unpublished data, 2018) in addition to another non-clinical pilot study which has been conducted among nursing home residents in Sandnes municipality (2).

A total of 25 women will be recruited based on the following inclusion criteria:

* More than 18 years of age
* Recurrent urinary tract infections (rUTI) (minimum of 2 episodes during the last 6 months, or minimum of 3 episodes during the last 12 months)
* Participants should be cooperative, capable of maintaining a patient diary, and providing urine samples according to a specified schedule

Exclusion criteria:

* Use of Hiprex during the last 6 months
* Regular use of aronia during the last 6 months
* Allergy to heat-treated aronia or apple
* Uncontrolled diabetes mellitus
* Use of blood-thinning medication (e.g. Warfarin, 'Marevan')

For recruitment of participants, information about the study will be posted on waiting room walls at Konsmo Doctors Office and through advertisement in local newspapers. Prior to study participation, written informed approval will be signed by all participants and they will be able to withdraw from the study at any time.

During the intervention period, study participants will consume 1 dL of the mixture every day for 6 months. This is equivalent to approximately half a breakfast glass of liquid. The aronia-mixture will preferably be consumed together with a meal or after finishing a meal. The mixture may be obtained in the fridge or in room temperature (but not heated), and study participants may consume the mixture in smaller portions throughout the day. Participants will be instructed to keep a patient diary and provide the following information:

* Deviations from the intervention protocol regarding the frequency and the dosage of aronia-mixture consumed.
* Observations regarding UTI symptoms should be described, i.e. symptoms of incipient infections, duration of symptoms, and when the symptoms cease. This applies to both untreated UTIs and medically treated infections.
* Other observations related to UTIs or intake of the aronia-mixture, i.e. changes in urine colour of urine, possible adverse effects, discomfort, etc.

For collection of urine samples, participants are provided with 10 items of 30 mL polypropylene tubes containing boric acid from the doctors office when entering the pilot study. More tubes will be provided if needed. The tubes will be labeled with date of delivery and names of study participants when delivering to the doctors office.

Urine samples for cultivation:

A urine sample will be collected by staff at the doctors office in Konsmo before the intervention period (pre-test). Additionally, a urine sample will be collected every time a urinary tract infection (UTI) is to be treated with antibiotics during the intervention period. De-identified samples will be sent for routine cultivation at Sorlandet Hospital by Dr. Ståle Tofteland and willl thereafter be routinely destroyed.

Urine samples for metabolite analysis:

30 mL urine samples will be collected by staff at the doctors office and sent for analysis of metabolites on day 0, 60, 120, and 180 of the intervention period. De-identified samples will be collected by Dr. Rune Slimestad who will also perform analysis continously after collection. The samples will be analyzed for phenolic metabolites using UHPLC-MS and quantified relative to urine concentration (creatinine). De-identified samples can be stored for up to 2 months in a freezer (-20 ℃) and then completely destroyed.

Data analysis:

The participants medical history of UTIs (12 months before initiation of the project and during the project period) will be obtained from the patients medical journals. Additionally, a patient diary from the project will provide information about transient, untreated infections, asymptomatic UTIs, other comments regarding the infection course, or intervention drinks.

The analysis work will focus on the main outcome measures and calculate dropouts from the study, changes in the frequency of treated (and untreated) UTIs, and changes in metabotyping.

1. Jurikova T et al. (2017) Fruits of Black Chokeberry Aronia melanocarpa in the Prevention of Chronic Diseases. Molecules;22(6).
2. Handeland, M. et al. (2014) Black chokeberry juice (Aronia melanocarpa) reduces incidences of urinary tract infection among nursing home residents in the long term - a pilot study. Nutr. Res. 34, 518-525.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Recurrent urinary tract infections (rUTI) (minimum of 2 episodes in the last 6 months, or minimum of 3 episodes in the last 12 months).
* Participants should be cooperative, capable of maintaining a patient diary, and providing urine samples according to a specified schedule.

Exclusion Criteria:

* Use of Hiprex in the last 6 months.
* Regular use of aronia in the last 6 months.
* Allergy to heat-treated aronia or apple.
* Uncontrolled diabetes mellitus.
* Use of blood-thinning medication (e.g. Warfarin).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The target group of the present study is females, as urinary tract infections are about 50 times more common in women than men. Thus, inclusion criteria is focusing on their biological sex and not their gender identity.
Enrollment: 23 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Study feasibility: recruitment of participants | From enrollment to end of treatment at 6 months
  Experiences related to the process of recruiting study participants
Study feasibility: drop-outs | From enrollment to end of treatment at 6 months
  Register the number of dropouts during the intervention period
Study feasibility: program adherence | From enrollment to end of treatment at 6 months
  Examine adherence to the program by study participants and staff
Study feasibility: duration of the intervention period | From enrollment to end of treatment at 6 months
  Acceptance of treatment duration among participants and recruiters

SECONDARY OUTCOMES:
Number of Urinary Tract Infections (UTIs) during the intervention period | From enrollment to end of treatment at 6 months
  Registration of the total number of symptomatic UTIs and symptom burden and antibiotic use prior to and during the intervention period. The results will contribute to establish power calculations required for a full-scale study (RCT).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Agder, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: No
According to ethical approval of the study protocol, we are not allowed to share individual participant data (IPD).